CLINICAL TRIAL: NCT01411332
Title: A Phase III Trial of Hypofractionated External Beam Image-Guided Highly Targeted Radiotherapy: The HEIGHT Trial
Brief Title: Hypofractionated Image-Guided Radiotherapy For Prostate Cancer: The HEIGHT Trial
Acronym: HEIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Alan Pollack, MD, PhD, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20100635
Record Dates: First submitted 2011-08-03; First posted 2011-08-08 (Estimated); Results first posted 2021-07-30 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm I: SIMRT (Active Comparator): 'Participants in this group will receive the Standard Fractionated Intensity Modulated Radiotherapy (SIMRT) consisting 40 fractions over 8 weeks.
  Interventions: Radiation: SIMRT
- Arm II: HTIMRT (Active Comparator): Participants in this group will receive the Hypofractionated Targeted Intensity Modulated Radiotherapy (HTIMRT) consisting of 38 fractions over 7.5 weeks.
  Interventions: Radiation: HTIMRT

INTERVENTIONS:
Radiation: SIMRT — A total dose of 80 Gy will be delivered in 40 fractions to the Clinical Target Volume (CTV).
  Other Names: Standard Fractionated Intensity Modulated Radiotherapy
  Arms: Arm I: SIMRT
Radiation: HTIMRT — Dose escalation to the Multiparametric MRI (MP-MRI) by dose painting at 2.35-2.40 Gy per fraction, while the rest of the Clinical Target Volume (CTV) receives 2.0 Gy a fraction to 76 Gy. The hypofractionated targeted (HT) boost region will receive an absolute dose of 89.3-91.2 Gy. Assuming an α/β ratio of 3.0, this would be equivalent to 95.5 Gy in 2.0 Gy fractions.
  Other Names: Hypofractionated Targeted Intensity Modulated Radiotherapy
  Arms: Arm II: HTIMRT

SUMMARY:
1. Delivery of directed hypofractionated targeted (HT) radiotherapy (RT) tumor boost to the dominant tumor lesion in the prostate as identified by multiparametric MRI will increase tumor eradication from the prostate.
2. Biomarker expression levels differ in the multiparametric MRI defined regions at high risk of harboring tumors that determine outcome.
3. 10-15% of men undergoing RT have Circulating DNA or tumor cells (CTC) that are related to an adverse treatment outcome.
4. Quality of life will not differ significantly between the treatment arms.
5. Prostate cancer-related anxiety will be reduced in the HTIMRT arm, because the patients will be aware that the dominant tumor will be targeted with higher radiation dose.

ELIGIBILITY:
Inclusion Criteria:

* A. Biopsy confirmed adenocarcinoma of the prostate.
* B. T1-T3a disease based on digital rectal exam.

  1. T1a is permitted if peripheral zone biopsies are positive.
  2. T3a disease based on MRI is acceptable.
* C. No evidence of metastasis by any clinical criteria or available radiographic tests.
* D. Gleason score 6-8.
* E. Patients with Gleason score 8 must be offered long term androgen deprivation therapy (ADT) and refuse such treatment because only 4-6 (±2 months) months (short term ADT) is permitted on this protocol. Gleason score ≥ 8 patients should be recommended to receive short term ADT in conjunction with RT. When given, the ADT recommended to begin after fiducial marker placement, if applicable; however, ADT is permitted to have been started up to two months prior to the signing of consent.

  1. Patients with Gleason score 8 disease must have <40 of the diagnostic tumor tissue involved with tumor.
  2. Patients with Gleason score ≤7 may be treated with 4-6 (±2 months) months of ADT.
* F. PSA ≤100 ng/mL within 3 months of enrollment. If PSA was above 100 and dropped to ≤100 with antibiotics, this is acceptable for enrollment.
* G. If PSA is >15 ng/ml or there is ≥ Gleason 8 disease, a bone scan should be obtained ≤4 months before enrollment and should be without evidence of metastasis. A questionable bone scan is acceptable if plain x-rays, CT and/or MRI are negative for metastasis.
* H. No previous pelvic radiotherapy
* I. No previous history of radical/total prostatectomy (suprapubic prostatectomy is acceptable)
* J. No concurrent, active malignancy, other than nonmetastatic skin cancer or early stage chronic lymphocytic leukemia (well-differentiated small cell lymphocytic lymphoma). If a prior malignancy is in remission for ≥ 5 years then the patient is eligible.
* K. Identifiable multiparameter functional MRI defined tumor lesion or lesions using a 1.5T or 3.0T MRI (3.0T preferable), that total in volume <33% of the prostate within 3 months prior to enrollment.

  a. Multiparametric functional including diffusion weighted imaging (DWI) of prostate and pelvis is required prior to protocol consideration
* L. Ability to understand and the willingness to sign a written informed consent document
* M. Zubrod performance status <2 (Karnofsky or Eastern Cooperative Oncology Group (ECOG) performance status may be used to estimate Zubrod)
* N. Willingness to fill out quality of life/psychosocial forms.
* O. Age ≥35 and ≤85 years.
* P. Serum testosterone is within 40% of normal assay limits (e.g., x=0.4*lower assay limit and x=.04*upper assay limit + upper assay limit),, taken within 4 months of enrollment. Patients who have been started on ADT prior to signing consent are not required to have a serum testosterone at this level prior to signing consent; but, a serum testosterone prior to fiducial marker placement is recommended.
* Q. Serum liver function tests (LFTs) taken within 3 months of enrollment.
* R. Complete blood counts taken within 3 months of enrollment.

Exclusion Criteria

* A. Previous pelvic radiotherapy.
* B. Previous history of radical prostatectomy.
* C. Concurrent, active malignancy, which is not nonmetastatic skin cancer or early stage chronic lymphocytic leukemia (well-differentiated small cell lymphocytic lymphoma). If a prior malignancy is in remission for < 5 years then the patient is not eligible
* D. Not willing to fill out quality of life/psychosocial questionnaires.

Ages: 35 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Pollack, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only 9 participants in Arm I and 7 participants in Arm II received study intervention.
Groups:
- Arm II: HTIMRT: All participants in this group will receive the Hypofractionated Targeted Intensity Modulated Radiotherapy (HTIMRT) consisting of a total of 38 fractions over 7.5 weeks.
  HTIMRT: Dose escalation to the Multiparametric MRI (MP-MRI) by dose painting at 2.35-2.40 Gy per fraction, while the rest of the Clinical Target Volume (CTV) receives 2.0 Gy a fraction to 76 Gy. The hypofractionated targeted (HT) boost region will receive an absolute dose of 89.3-91.2 Gy. Assuming an α/β ratio of 3.0, this would be equivalent to 95.5 Gy in 2.0 Gy fractions.
Period: Enrollment
Arm/Group | Arm I: SIMRT | Arm II: HTIMRT
Started | 9 | 9
Completed | 9 | 7
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Treatment
Arm/Group | Arm I: SIMRT | Arm II: HTIMRT
Started | 9 | 7
Completed | 8 | 7
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: SIMRT | Arm II: HTIMRT | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 8 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biopsy Failure
Description: Number of participants showing positive prostate biopsy finding post treatment.
Time Frame: Up to 2.25 years
Population: Of the 18 enrolled participants, only 16 participants were still enrolled at the 2.25 years follow up. Of the 16 participants, only 9 participants were able to complete the post treatment biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: SIMRT | Arm II: HTIMRT
Number analyzed (Participants) | 4 | 5
Participants | 0 | 2

2. Secondary Outcome: Toxicity Rate
Description: Toxicity rate will be reported as the number of participants experiencing any treatment-related adverse events. Acute and Late Toxicity will be evaluated by treating physician using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0. Acute toxicity will be defined as any treatment-related adverse event during and within 3 months of completing treatment. Late Toxicity will be defined as any treatment-related adverse events occurring more than 3 months after treatment completion.
Time Frame: Up to 6 years
Population: Only 16 participants received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: SIMRT | Arm II: HTIMRT
Number analyzed (Participants) | 9 | 7
Participants
  Treatment-related Serious Adverse Events (SAEs) | 1 | 0
  Treatment-related Acute Toxicity (<=3 months of completing treatment) | 9 | 7
  Treatment-related Grade 3 or higher Acute Toxicity | 0 | 0
  Treatment-related Late Toxicity (>3 months after completing treatment) | 7 | 5
  Treatment-related Grade 3 or higher Late Toxicity | 1 | 0

3. Secondary Outcome: Mortality
Description: Mortality will be reported as overall survival and failure free survival. Overall survival is defined as the elapsed time from start of radiotherapy to death from any cause. Failure free survival is defined as the elapsed time from start of radiotherapy to first documented evidence of biochemical or clinical failure or death from any cause, whichever occurs first. In the absence of any event defining failure, follow-up time will be censored at the date of last documented failure-free status.
Time Frame: Up to 6 years
Population: Only 16 participants received study intervention.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Arm I: SIMRT | Arm II: HTIMRT
Number analyzed (Participants) | 9 | 7
months
  Failure Free Survival | 64.9 [64.8 to 65.6] | 65.0 [64.1 to 65.6]
  Overall Survival | 64.9 [64.8 to 65.6] | 65.0 [64.1 to 65.6]

4. Secondary Outcome: Failure Rate
Description: Failure rate will be reported as the incidence of biochemical or clinical failure. Biochemical failure is defined is an increase of 2 or greater from nadir of Prostate Specific Antigen (PSA) levels. Clinical Failure is defined as newly identified extension outside the prostate after initial regression, or urinary obstructive symptoms with carcinoma or regional/distant failure due to radiographic evidence metastasis.
Time Frame: Up to 6 years
Population: Only 16 participants received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: SIMRT | Arm II: HTIMRT
Number analyzed (Participants) | 9 | 7
Participants
  Biochemical Failure | 0 | 0
  Clinical Failure | 0 | 0

5. Secondary Outcome: EPIC SF-12 Scores
Description: Health-related Quality of Life (HRQOL) will be measured using the Expanded Prostate Cancer Index Composite and Medical Outcomes Study SF-12 (EPIC SF-12) to evaluate patient function and satisfaction after prostate cancer treatment. Response options for each item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better HRQOL.
Time Frame: At baseline, at last week of treatment (Up to 8 weeks), at 6 weeks after treatment (Up to 14 weeks), at 3 months after treatment (Up to 20 weeks), at 9 months after treatment (Up to 44 weeks).
Population: Only 16 participants received study intervention. Not all participants completed the survey at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I: SIMRT | Arm II: HTIMRT
Number analyzed (Participants) | 9 | 7
score on a scale
  Urinary Function (Incontinence): Baseline (Prior to treatment) | 90.8 (14.2) | 89.3 (15.7)
  Urinary Function (Incontinence): Last week of treatment (Up to 8 weeks) | 82.2 (23.9) | 84.8 (27.1)
  Urinary Function (Incontinence): 6 weeks after treatment (Up to 14 weeks) | 87.3 (14.0) | 82.1 (24.5)
  Urinary Function (Incontinence): 3 months after treatment (Up to 20 weeks) | 93.8 (10.8) | 93.2 (12.8)
  Urinary Function (Incontinence): 9 months after treatment (Up to 44 weeks): number analyzed (Participants) | 8 | 5
  Urinary Function (Incontinence): 9 months after treatment (Up to 44 weeks) | 88.8 (12.0) | 83.8 (15.2)
  Urinary Symptoms (Irritative/Obstructive): Baseline (Prior to treatment) | 92.1 (5) | 82.1 (19.5)
  Urinary Symptoms (Irritative/Obstructive): Last week of treatment (Up to 8 weeks) | 81.1 (17.6) | 73.6 (25.6)
  Urinary Symptoms (Irritative/Obstructive): 6 weeks after treatment (Up to 14 weeks) | 91.5 (7.9) | 82.1 (22.9)
  Urinary Irritative/Obstructive: 3 months after treatment (Up to 20 weeks) | 93.3 (12) | 89.3 (12.4)
  Urinary Irritative/Obstructive: 9 months after treatment (Up to 44 weeks): number analyzed (Participants) | 8 | 5
  Urinary Irritative/Obstructive: 9 months after treatment (Up to 44 weeks) | 95.6 (5.6) | 79 (16)
  Bowel Habits: Baseline (Prior to treatment): number analyzed (Participants) | 8 | 7
  Bowel Habits: Baseline (Prior to treatment) | 94.3 (6.3) | 88.7 (15.9)
  Bowel Habits: Last week of treatment (Up to 8 weeks) | 90.3 (13.7) | 92.3 (5.6)
  Bowel Habits: 6 weeks after treatment (Up to 14 weeks): number analyzed (Participants) | 8 | 7
  Bowel Habits: 6 weeks after treatment (Up to 14 weeks) | 98.4 (2.2) | 94 (6.7)
  Bowel Habits: 3 months after treatment (Up to 20 weeks) | 95.8 (7.5) | 96.4 (4.5)
  Bowel Habits: 9 months after treatment (Up to 44 weeks): number analyzed (Participants) | 8 | 4
  Bowel Habits: 9 months after treatment (Up to 44 weeks) | 93.8 (8) | 86.5 (9.2)
  Sexual Function: Baseline (Prior to treatment): number analyzed (Participants) | 9 | 6
  Sexual Function: Baseline (Prior to treatment) | 49.4 (29.2) | 37.5 (32.7)
  Sexual Function: Last week of treatment (Up to 8 weeks): number analyzed (Participants) | 9 | 6
  Sexual Function: Last week of treatment (Up to 8 weeks) | 41.5 (29.6) | 35.9 (30.1)
  Sexual Function: 6 weeks after treatment (Up to 14 weeks): number analyzed (Participants) | 9 | 6
  Sexual Function: 6 weeks after treatment (Up to 14 weeks) | 43.8 (27.3) | 33.6 (31.2)
  Sexual Function: 3 months after treatment (Up to 20 weeks): number analyzed (Participants) | 8 | 7
  Sexual Function: 3 months after treatment (Up to 20 weeks) | 35.1 (22.1) | 40.3 (37.9)
  Sexual Function: 9 months after treatment (Up to 44 weeks): number analyzed (Participants) | 8 | 4
  Sexual Function: 9 months after treatment (Up to 44 weeks) | 28 (14.9) | 44.8 (40)
  Hormonal Function: Baseline (Prior to treatment): number analyzed (Participants) | 8 | 7
  Hormonal Function: Baseline (Prior to treatment) | 88.8 (11.9) | 77.9 (25.3)
  Hormonal Function: Last week of treatment (Up to 8 weeks) | 90 (10.9) | 79.3 (25.6)
  Hormonal Function: 6 weeks after treatment (Up to 14 weeks) | 84.4 (14.9) | 71.4 (18.2)
  Hormonal Function: 3 months after treatment (Up to 20 weeks): number analyzed (Participants) | 8 | 7
  Hormonal Function: 3 months after treatment (Up to 20 weeks) | 89.4 (16.8) | 79.3 (16.4)
  Hormonal Function: 9 months after treatment (Up to 44 weeks): number analyzed (Participants) | 8 | 5
  Hormonal Function: 9 months after treatment (Up to 44 weeks) | 91.9 (11.3) | 83 (14.4)

6. Secondary Outcome: MAX-PC Scores
Description: Health-related quality of life (HRQOL) will be measured using the scores on the Modified 18-item Memorial Anxiety Scale for Prostate Cancer (MAX-PC). The scale consists of 18 items (e.g. "I thought about prostate cancer even though I didn't mean to.") scored on a scale from 0 ("not at all") to 3 ("often"). Total scores range from 0 to 54, with higher scores indicating higher levels of anxiety.
Time Frame: as for outcome 5
Population: Only 16 participants received study intervention. Not all participants completed the survey at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I: SIMRT | Arm II: HTIMRT
Number analyzed (Participants) | 9 | 7
score on a scale
  Baseline (Prior to treatment) | 10.6 (9.0) | 16.6 (9.2)
  Last week of treatment (Up to 8 weeks): number analyzed (Participants) | 8 | 7
  Last week of treatment (Up to 8 weeks) | 12.3 (7.7) | 13.9 (7.9)
  6 weeks after treatment (Up to 14 weeks) | 12.9 (3.3) | 13.0 (8.1)
  3 months after treatment (Up to 20 weeks) | 10.6 (5.0) | 11.3 (3.5)
  9 months after treatment (Up to 44 weeks): number analyzed (Participants) | 8 | 5
  9 months after treatment (Up to 44 weeks) | 10.0 (6.8) | 9.6 (1.5)

7. Secondary Outcome: Biomarker Expression in Prostate Tumor Regions
Description: The amount of biomarker expression will be evaluated via immunohistochemistry (IHC) from ultrasound guided prostate biopsy tissue samples for both functional MRI suspicious regions and those that are not suspicious.
Time Frame: Up to 3 years
Population: While tissue was collected for biomarker, none of the samples were analyzed because of insufficient patient numbers and power to draw conclusions. These types of analyses are done in batches and we never reached an appropriate threshold of cases to perform even exploratory analyses. No samples have been analyzed for biomarkers using IHC.
Arm/Group | Arm I: SIMRT | Arm II: HTIMRT
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Incidence of Circulating Free DNA
Description: Incidence of circulating free DNA, as assessed from blood samples.
Time Frame: Up to 3 years
Population: While blood was collected for cfDNA assessment, none of the samples were analyzed because of insufficient patient numbers and power to draw conclusions. These types of analyses are done in batches and we never reached an appropriate threshold of cases to perform even exploratory analyses. No samples have been analyzed for cfDNA.
Arm/Group | Arm I: SIMRT | Arm II: HTIMRT
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 years
Arm/Group | Arm I: SIMRT | Arm II: HTIMRT
All-Cause Mortality (participants affected / at risk) | 0/9 | 1/7
Serious Adverse Events (participants affected / at risk) | 2/9 | 3/7
Other Adverse Events (participants affected / at risk) | 9/9 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: SIMRT (N=9) | Arm II: HTIMRT (N=7)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: SIMRT (N=9) | Arm II: HTIMRT (N=7)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 8 (15) | 6 (6)
Depression (Psychiatric disorders) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 7 (15) | 2 (4)
Edema Limbs (General disorders) | 1 (2) | 4 (4)
Ejaculation Disorder (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Low Testosterone (Endocrine disorders) | 1 (1) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 4 (4) | 3 (6)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Fatigue (General disorders) | 5 (5) | 6 (9)
Fecal Incontinence (Gastrointestinal disorders) | 0 (0) | 2 (3)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Blood on Rectum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hard Stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (4) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hot Flashes (Vascular disorders) | 1 (1) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Low Testosterone (Investigations) | 1 (1) | 1 (1)
Libido decreased (Psychiatric disorders) | 2 (2) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1) | 1 (1) — Testicular tenderness
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (2) | 1 (1)
Prostatic Obstruction (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Rectal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Renal and Urinary Disorder - Other (Renal and urinary disorders) | 1 (1) | 0 (0)
Low Testosterone (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular Disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Atrophic testicle
Testicular Disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Decreased Testosterone Level
Testicular Pain (Reproductive system and breast disorders) | 1 (1) | 1 (2)
Urinary Frequency (Renal and urinary disorders) | 7 (19) | 7 (10)
Urinary Incontinence (Renal and urinary disorders) | 6 (11) | 3 (5)
Urinary Retention (Renal and urinary disorders) | 4 (8) | 3 (6)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Tract Pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Urgency (Renal and urinary disorders) | 9 (21) | 6 (12)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Polycitemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest Pain - Cardiac (Cardiac disorders) | 1 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Creatinine Increased (Investigations) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (6) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 2 (2)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Irritated Seborrheic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Right knee pain
Penile Infection (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Squamous Cell Carcinoma in SITU Bowens Disease (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight gain (Investigations) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT01411332/Prot_SAP_000.pdf